CLINICAL TRIAL: NCT02007629
Title: An Open-label, International, Multicenter, Single-arm, Uncontrolled, Phase IIIb Study of Riociguat in Patients With Pulmonary Arterial Hypertension (PAH) Who Demonstrate an Insufficient Response to Treatment With Phosphodiesterase-5 Inhibitors (PDE-5i)
Brief Title: Riociguat Clinical Effects Studied in Patients With Insufficient Treatment Response to Phosphodiesterase-5 Inhibitor
Acronym: RESPITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16719; 2013-001759-10 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2018-12

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riociguat (Experimental): Subjects received riociguat film coated immediate-release (IR) tablet 3 times a day (tid) with or without food at a starting dose of 1.0 milligram (mg) and increased by 0.5 mg increments at 2-weekly intervals to a maximum of 2.5 mg tid, until Week 8 (titration phase). An optimal dose was determined based on systolic blood pressure (SBP) and well-being. Thereafter, riociguat continued at the optimal individual dose until Week 24 (Main phase). Dose reductions or stop of study medication for safety reasons were allowed at any time. Increases or re-increases in 0.5 mg steps (maximum dose 2.5 mg) were possible at the investigator's discretion weighing the benefit with potential risks implied. Subjects were offered participation in EDSP and received riociguat 2.5 mg film coated IR tablet 3 tid with or without food for 18 months or until reimbursement.
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Riociguat / BAY63-2521 film-coated tablets will be used in this study at a dosage of either 0.5, 1.0, 1.5, 2.0, and 2.5 mg. 3 times daily

SUMMARY:
BAY63-2521 Riociguat leads to the relaxation of smooth muscle cells in pulmonary arteria and may also inhibit abnormal remodeling of lung blood vessels. In patients with pulmonary arterial hypertension Riociguat showed to reduce the pulmonary blood pressure and improved the right heart function without unacceptable side effects. Here dose of Riociguat will be adjusted over 8 weeks then a Maintenance Phase of 16 weeks follows. Patients with Pulmonary Arterial Hypertension treated with stable doses of Phosphodiesterase Type-5 Inhibitors (Eg Sildenafil, Tadalafil) not appropriately responding to therapy will be included. Based on previous evidence and on the different modes of action an improvement of exercise capacity, heart function and quality of life may be expected if PDE5i treatment is transitioned to riociguat.

Where Riociguat is pending market approval or reimbursement once the treatment phase is completed drug can be made available for another 18 months (Extended Drug Supply Phase - EDSP) under study conditions. Patients may also transition at the end of the maintenance period or any time during the EDSP to any program that is intended to provide riociguat until drug approval/reimbursement, e.g. a long-term extension study, compassionate use or named patient program. Study termination is also possible at any time.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (18 -75 years of age) with idiopathic, familial, drug/toxin induced and associated PAH due to congenital heart disease (Group I / Dana Point Classification of PH) demonstrating insufficient response to treatment with PDE-5i for at least 3 months
* Patients with and without endothelin receptor antagonist (ERA) therapy
* World Health Organization Functional Class (WHO FC) III at screening
* 6-minute walking distance (6MWD) of 165-440 m
* Cardiac index <3.0 L/min/m*2.

Exclusion Criteria:

* All types of PH except subtypes of Dana Point Group I specified in the inclusion criteria
* Evidence of clinically significant restrictive or obstructive parenchymal lung diseases
* Diffusing capacity of the lung for carbon monoxide (DLCO) <30% predicted
* History or active state of serious hemoptysis / pulmonary hemorrhage including those managed by bronchial artery embolization
* Patients unable to perform a valid 6MWD test
* Pregnant women (i.e. positive pregnancy test or other signs of pregnancy), or breast feeding women, or women with childbearing potential not using a combination of 2 effective methods of birth control, for example a combination of condoms with a safe and highly effective contraception method (prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device) or a double barrier method is used throughout the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-02-18; Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 6 Minute Walking Distance (6MWD) | Baseline, Week 12 and Week 24
  6MWD test was used to measure the subjects functional exercise capacity. Subjects were instructed to walk alone, not run, from one end to the other end of the walking course, at their own pace, while attempting to cover as much ground as possible in 6 minutes. No "warm-up" period was performed before the test. Investigators have not walked with the subjects. This was an encouraged test (the person conducting the test encouraged subjects to walk farther or faster by using only standardized phrases).

OTHER OUTCOMES:
Change From Baseline in Cardiac Index | Baseline, Week 24
  The cardiac output was measured by using the thermodilution methodology and a respective electronic device. The cardiac index was assessed by dividing the cardiac output by the person's BSA.
Change From Pre-treatment in N-Terminal Pro-Brain Natriuretic Peptide (NTproBNP) | Baseline, Week 12 and Week 24
  NT-proBNP cardiac biomarker was used to detect, diagnose, and evaluate the severity of heart failure. A higher level of the marker was indicative of heart failure.
Change From Baseline in World Health Organization Functional Class (WHO FC) | Baseline, Week 12 and Week 24
  WHO FC assessment of PAH ranged from functional class I (subjects with PH but without resulting limitation of physical activity); class II (subjects with PH resulting in slight limitation of physical activity); class III (subjects with PH resulting in marked limitation of physical activity); class IV (subjects with PH with inability to carry out any physical activity without symptoms); and class V death. Changes to a lower WHO FC resemble improvement; changes to a higher functional class resemble deterioration of PAH.
Percentage of Subjects With Clinical Worsening | Baseline to Week 24
  Clinical worsening was defined as death (all-cause mortality); atrial septostomy; lung transplantation; non-planned PAH-related hospitalisation; start of new PAH treatment (ERA, inhaled or oral prostanoid) or modification of pre-existing treatment, initiation of intravenous or subcutaneous prostanoids; persistent decrease of greater than (>) 15% from baseline or >30% from last measurement in 6MWD; persistent worsening of WHO FC; or appearance or worsening of signs/symptoms of right heart failure not responding to optimised oral diuretic therapy. All identified and suspected clinical worsening events were confirmed by independent central adjudication.
Change From Baseline in European Quality of life (Qol)-Group (EQ)-5D Questionnaire | Baseline, Week 12 and Week 24
  EQ-5D was a standardized instrument which was used to measure the health outcome. The EQ-5D was a selfreport questionnaire and needed to be completed by the subject. After the subject filled in the questionnaire, the questionnaire was transferred into the electronic case report form (eCRF). EQ-5D was calculated by two types of questionnaires Part A (descriptive health profile) and Part B (visual analogue scale). Part A, EQ-5D comprised 5-item questionnaires to measure own health profile status (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each measure has three levels (1. no problems, 2. some problems, 3. extreme problems). In Part B, visual analogue rating scale to measure how good or bad a health state was. Scale was drawn by using thermometer-like scale, on which the best state imagine was marked as 100 and worst state imagine was marked as 0.
Change from pre-treatment of 6MWD | Baseline, Week 12 and Week 24
Percentage of Subjects Without Clinical Worsening who Achieve at Least WHO FC II and an Improvement in 6 MWD of Greater Than or Equal to (>=) 30 meters | Baseline, Week 12 and Week 24
  Percentage of subjects without clinical worsening who achieve at least who FC II and an improvement in 6 MWD of >= 30 meters were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (26):
- United States (7):
  - La Jolla, California
  - Sacramento, California
  - Iowa City, Iowa
  - Boston, Massachusetts
  - St Louis, Missouri
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Montreal, Quebec, Canada
- Prague, Czechia
- France (3):
  - Grenoble
  - Le Kremlin-Bicêtre
  - Marseille
- Germany (6):
  - Heidelberg, Baden-Wurttemberg
  - Regensburg, Bavaria
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
- Italy (2):
  - Rome, Lazio
  - Pavia, Lombardy
- Zurich, Switzerland
- United Kingdom (3):
  - Newcastle upon Tyne, Tyne and Wear
  - Clydebank, West Dunbartonshire
  - London

REFERENCES:
- [Result] Hoeper MM, Klinger JR, Benza RL, Simonneau G, Langleben D, Naeije R, Corris PA. Rationale and study design of RESPITE: An open-label, phase 3b study of riociguat in patients with pulmonary arterial hypertension who demonstrate an insufficient response to treatment with phosphodiesterase-5 inhibitors. Respir Med. 2017 Jan;122 Suppl 1:S18-S22. doi: 10.1016/j.rmed.2016.11.001. Epub 2016 Nov 5. PMID 27887774
- [Result] Hoeper MM, Simonneau G, Corris PA, Ghofrani HA, Klinger JR, Langleben D, Naeije R, Jansa P, Rosenkranz S, Scelsi L, Grunig E, Vizza CD, Chang M, Colorado P, Meier C, Busse D, Benza RL. RESPITE: switching to riociguat in pulmonary arterial hypertension patients with inadequate response to phosphodiesterase-5 inhibitors. Eur Respir J. 2017 Sep 9;50(3):1602425. doi: 10.1183/13993003.02425-2016. Print 2017 Sep. PMID 28889107
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/